CLINICAL TRIAL: NCT02267577
Title: Accuracy Assessment of an Automatic Blood Pressure Measurement Device in Adult Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Marsh Rice University (Other)
Responsible Party: Principal Investigator, Rebecca Richards-Kortum, Stanley C. Moore Professor of Bioengineering, William Marsh Rice University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 14-082F-A; 51262 (Other Grant/Funding Number: Merck for Mothers: 51262)
Record Dates: First submitted 2014-10-09; First posted 2014-10-17 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Pre Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Participants enrolled in the study will have their blood pressure measured multiple times with both the GE Dinamap Procare commercial blood pressure monitor and Sphygmo, the experimental blood pressure monitoring device.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Adults Volunteers (Experimental): Men and women over the age of 18 will have their blood pressure measured with both the Sphygmo: Automatic Blood Pressure Monitor device and the GE Dinamap ProCare automatic blood pressure monitor.
  Interventions: Device: Sphygmo: Automatic Blood Pressure Monitor; Device: GE Dinamap ProCare Automatic Blood Pressure Monitor

INTERVENTIONS:
Device: Sphygmo: Automatic Blood Pressure Monitor — A team of engineers from Rice University has recently developed Sphygmo, an ambulatory, low-cost blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals.
Device: GE Dinamap ProCare Automatic Blood Pressure Monitor — This commercially available gold standard blood pressure monitor will be used as a control to assess the accuracy of the Sphygmo device.

SUMMARY:
The research team has developed an automatic blood pressure monitor (Sphygmo) to be used for the monitoring and diagnosis of pre-eclampsia in pregnant women, particularly in low-resource settings where current monitoring is limited.

90 adult volunteers will be enrolled by researchers at Rice University. The participant will be seated in a comfortable chair with arm at heart level. Arm circumference will be measured and a blood pressure cuff will be placed on the arm. The cuff will be inflated and blood pressure measurements will be taken by a commercially available device and by the Sphygmo device. Blood pressure measurements from both devices will be recorded. The participant's blood pressure will be measured up to 9 times with a waiting period of 45-60 seconds between each measurement.

The results of this study will be used to optimize the blood pressure detection algorithm and thus further develop the device.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Willing and able to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2017-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R Kortum, PhD, Principal Investigator — William Marsh Rice University
Locations (1):
- Rice University, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adult Volunteers: Men and women over the age of 18 who will have their blood pressure measured using both the experimental blood pressure monitor (Sphygmo), and the gold-standard, commercial blood pressure monitor (GE Dinamap ProCare).
Period: Overall Study
Arm/Group | Healthy Adult Volunteers
Started | 85
Completed | 81
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Adults Volunteers: Men and women over the age of 18
  Sphygmo: Automatic Blood Pressure Monitor: A team of engineers from Rice University has recently developed Sphygmo, an ambulatory, low-cost blood pressure monitor for use in the diagnosis and management of pre-eclampsia in low-resource hospitals.
Arm/Group | Adults Volunteers
Number analyzed (Participants) | 85
Age, Continuous [Median (Full Range); unit: years] | 50 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Blood Pressure Measurement by Sphygmo Relative to the Clinical Standard.
Description: Mean difference of systolic and diastolic blood pressure readings between Sphygmo device and the gold standard sphygmomanometer.
Time Frame: Blood pressure was measured an average of 9 times for each participant during their single visit and the mean of these measurements was recorded and used for analysis. The measurement period lasted approximately 30-45 minutes.
Population: Data from nine participants of the original 81 who completed the study was excluded on account of the observer reporting a difficulty in hearing, movement, or uncertainty with the measurement.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Healthy Adult Volunteers: Men and women over the age of 18 who had their blood pressure measured using both the experimental device (Sphygmo) as well as the commercial, gold-standard monitor (GE Dinamap ProCare).
Arm/Group | Healthy Adult Volunteers
Number analyzed (Participants) | 72
mmHg
  Mean Systolic BP - Sphygmo | 122.5 (14.9)
  Mean Diastolic BP Difference - Sphygmo | 74.5 (11.1)
  Mean Systolic BP - GE Dinamap | 123.1 (17.7)
  Mean Diastolic BP - GE Dinamap | 72.1 (12.6)

2. Primary Outcome: Percentage of Sphygmo Readings That Were With < 5 mmHg, < 10 mmHg, and < 15 mmHg of the Readings by the Gold Standard Sphygmomanometer.
Description: The British Hypertension society defines a specific criteria for the accuracy of a sphygmomanometer. Devices are graded according to the cumulative percentage of readings that have an absolute difference between the more favorable observer's mercury sphygmomanometer readings and the test device of < 5 mmHg, < 10 mmHg, and < 15 mmHg. A letter grade of "A" requires that over 60%, 85%, and 95% were achieved in the < 5 mmHg, < 10 mmHg, and <15 mmHg categories, respectively. A letter grade of "B" requires that over 50%, 75%, and 90% were achieved in the < 5 mmHg, < 10 mmHg, and <15 mmHg categories, respectively. The test device achieved a grade of (B/B) with the validation data from this study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of measurements in that range
Groups:
- Adults Volunteers: Men and women over the age of 18 who will have their blood pressure measured using both the experimental blood pressure monitor (Sphygmo), and the gold-standard, commercial blood pressure monitor (GE Dinamap ProCare).
Arm/Group | Adults Volunteers
Number analyzed (Participants) | 72
percentage of measurements in that range
  Systolic Difference <5 mmHg | 56
  Systolic Difference <10 mmHg | 79
  Systolic Difference <15 mmHg | 92
  Diastolic Difference <5 mmHg | 53
  Diastolic Difference <10 mmHg | 77
  Diastolic Difference <15 mmHg | 90

ADVERSE EVENTS:
Arm/Group | Adults Volunteers
Serious Adverse Events (participants affected / at risk) | 1/85
Other Adverse Events (participants affected / at risk) | 0/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults Volunteers (N=85)
High Blood Pressure (Cardiac disorders) | 1 (1) — One healthy volunteer presented with abnormally high blood pressure. EMS was called and the subject was evaluated. Following the evaluation, the subject was advised to visit their primary care physician regarding their high blood pressure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No